CLINICAL TRIAL: NCT00696085
Title: Prevention of Fetal Alcohol Damage Using Maternal Blood Markers
Brief Title: Fetal Alcohol Damage Prevention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Lewis B. Holmes, M.D., Chief, Genetics Unit, MassGeneral Hospital for Children
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1999-P-008236/21
Record Dates: First submitted 2008-06-06; First posted 2008-06-12 (Estimated); Last update posted 2008-06-12 (Estimated); Status verified 2008-06

CONDITIONS: Fetal Alcohol Syndrome; Substance Abuse
Keywords: fetal alcohol exposure; blood markers of alcohol use; brief intervention
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders; Substance-Related Disorders | interventions — Crisis Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- I (Other): Pregnant women are recruited and screened for alcohol use using a validated alcoholism screening questionnaire. Those who screen positive are then entered into the next phase of the study.
  Interventions: Behavioral: Brief motivational intervention

INTERVENTIONS:
Behavioral: Brief motivational intervention — The women who have positive alcohol screening questionnaires and a random sample of women who screen negative are entered into the next phase of the study. They have blood drawn for the markers of alcohol use, are told of the results and are given brief intervention about alcohol use.
  Other Names: Motivational Intervention; Brief Intervention

SUMMARY:
The goal of this study was to determine whether a series of blood markers of alcohol use obtained from alcohol using pregnant women could help them to change their behavior.

DETAILED DESCRIPTION:
This study involved screening pregnant women with an alcoholism screening questionnaire and obtaining blood from those women who screened positive and a subset of women who screened negative. Each woman who had blood drawn were informed of their results, educated about alcohol use in pregnancy and had a brief intervention about their alcohol use, if appropriate. They were monitored throughout the pregnancy with additional blood tests obtained, depending upon their stage in pregnancy. After birth the babies were examined for any signs of alcohol exposure.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women seen at one of the obstetric clinics in the study and willing to give a blood sample

Exclusion Criteria:

* over 36 week gestation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 612 (Actual)
Dates: Start 2004-03; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Decrease in drinking | during the pregnancy

SECONDARY OUTCOMES:
improved infant size | after pregnancy finished

CONTACTS AND LOCATIONS:
Overall Officials: Lewis B Holmes, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States